CLINICAL TRIAL: NCT01911078
Title: Renal Sympathetic Denervation in Metabolic Syndrome (Metabolic Syndrome Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CI-12-079-EU-RD
Record Dates: First submitted 2013-07-24; First posted 2013-07-30 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic syndrome; Renal denervation; Renal artery; Muscle sympathetic nerve activity
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Renal Denervation Group (Other): Subjects receiving renal denervation procedure.
  Interventions: Procedure: Renal Denervation; Device: EnligHTN™ Renal Denervation System.
- Control Group (No Intervention): Subjects not receiving renal denervation procedure.
  Subjects are randomized in a 3:1 ratio to either Renal Denervation Group or Control Group.

INTERVENTIONS:
Procedure: Renal Denervation — Renal artery ablation with the EnligHTN™ Renal Denervation System.
  Arms: Renal Denervation Group
Device: EnligHTN™ Renal Denervation System.
  Arms: Renal Denervation Group

SUMMARY:
The purpose of this clinical investigation is to determine the effects of renal sympathetic denervation on insulin resistance and muscle sympathetic nerve activity in patients with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patient with office blood pressure ≥140/90 mmHg and 24-hour ambulatory blood pressure ≥130/80 mmHg at Baseline despite the stable use of at least two anti-hypertensive drugs at maximum tolerated doses of the patient for at least 4 weeks
* Patient with a fasting glucose ≥100 mg/dL (≥5.6 mmol/L) at Baseline or on drug treatment for elevated glucose
* Patient with a waist circumference ≥102 cm (≥40 inches) for male or ≥88 cm (≥35 inches) for female at Baseline
* Patient with any of the remaining two metabolic syndrome diagnostic criteria listed as follows at Baseline

  * Triglycerides ≥150 mg/dL (≥1.7 mmol/L) or on drug treatment for elevated triglycerides
  * High density lipid cholesterol (HDL-C) <40 mg/dL (<1.03 mmol/L) for male or <50 mg/dL (<1.30 mmol/L) for female or on drug treatment for reduced HDL-C
* Patient is ≥18 and ≤70 years old
* Patient must be able and willing to provide written informed consent to participate in this clinical investigation
* Patient must be able and willing to comply with the required follow-up schedule

Exclusion Criteria:

* Patient with secondary hypertension
* Patient with type I diabetes mellitus or type II diabetes mellitus requiring insulin therapy
* Patient with prior renal angioplasty, renal denervation, indwelling renal stents and/or aortic stent grafts
* Patient with renal arteries <4.0 mm in diameter
* Patient with significant renovascular abnormalities (such as renal artery stenosis >30%)
* Patient with an estimated glomerular filtration rate (eGFR) of <45 mL/min per 1.73 m2 using the Modified Diet in Renal Disease (MDRD) formula
* Patient with hemodynamically significant valvular heart disease, as determined by Study Investigator
* Patient has had a myocardial infarction, unstable angina pectoris or cerebrovascular accident less than 180 days at Baseline or is expected to have cardiovascular intervention within the next 180 days
* Patient is in chronic atrial fibrillation/flutter or with severe conduction abnormalities or with an implantable cardioverter defibrillator (ICD) or pacemaker whose settings cannot allow for radiofrequency (RF) energy delivery
* Patient is currently being treated with drugs that cause salt retention (such as systemic corticosteroids or fludrocortisone), centrally acting sympatholytic antihypertensive drugs, direct vasodilators (such as alpha blockers) and continuous positive airway pressure (CPAP) therapy for obstructive sleep apnea
* Patient with an active systemic infection or blood-clotting abnormalities or allergy to radiographic contrast
* Patient is pregnant or of childbearing potential and is not using adequate contraceptive methods or nursing
* Patient is participating in another clinical investigation
* Patient has a life expectancy less than 12 months, as determined by Study Investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in insulin resistance from baseline to 3 months after renal denervation | Baseline and Month 3
  To determine the effects of renal sympathetic denervation on insulin resistance (determined by the Homeostasis Model Assessment - Insulin Resistance method) at 3 months after renal denervation
Change in muscle sympathetic nerve activity (MSNA) from baseline to 3 months after renal denervation | Baseline and Month 3
  To determine the effects of renal sympathetic denervation on MSNA at 3 months after renal denervation

SECONDARY OUTCOMES:
Change in insulin resistance from baseline to 12 months after renal denervation | Baseline and Month 12
  To determine the effects of renal sympathetic denervation on insulin resistance long-term (12 months after renal denervation).
Change in muscle sympathetic nerve activity (MSNA) from baseline to 12 months after renal denervation | Baseline and Month 12
  To determine the effects of renal sympathetic denervation on MSNA long-term (12 months after renal denervation).

CONTACTS AND LOCATIONS:
Locations (1):
- Hippocration Hospital, University of Athens, Athens, Greece